CLINICAL TRIAL: NCT02602470
Title: A Study of Patient Preferences and Drivers of Treatment Satisfaction in Patients With Rosacea
Brief Title: Preferences & Treatment Satisfaction Drivers in Rosacea Patients
Status: Completed | Type: Observational
Sponsor: LEO Pharma (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18575
Record Dates: First submitted 2015-11-10; First posted 2015-11-11 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2017-04

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rosacea treated patients: Patients using topical rosacea treatment
  Interventions: Drug: Azelaic Acid Gel including: Finacea (Azelaic Acid Gel 15%, BAY39-6251); Drug: Azelaic Acid Cream; Drug: Metronidazole gel; Drug: Metronidazole cream; Drug: Metronidazole Emulsion; Drug: Metronidazole Lotion; Drug: Brimonidine Tartrate Gel

INTERVENTIONS:
Drug: Azelaic Acid Gel including: Finacea (Azelaic Acid Gel 15%, BAY39-6251) — Azelaic Acid Gel 15%, Azelaic Acid Gel 15% w/Cleanser & Moisturizing
Drug: Azelaic Acid Cream — Azelaic Acid Cream 20%
Drug: Metronidazole gel — Metronidazole Gel 1%, Metronidazole Gel 1% w/ Cleanser, Metronidazole Gel 0.75%, Metronidazole Gel 0.75% w/ Cleanser
Drug: Metronidazole cream — Metronidazole Cream 1%, Metronidazole Cream 0.75%, Metronidazole Cream 0.75% w/ Cleanser
Drug: Metronidazole Emulsion — Metronidazole Emulsion 0.75%
Drug: Metronidazole Lotion — Metronidazole Lotion 0,75%
Drug: Brimonidine Tartrate Gel — Brimonidine Tartrate Gel 0.33%

SUMMARY:
To survey patients with rosacea about their rosacea treatment preferences as well as to assess potential drivers of rosacea treatment satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of at least 18 years of age at index date
* At least one prescription for a topical rosacea treatments: Azelaic Acid Gel, Azelaic Acid Cream, Metronidazole Gel, Metronidazole Cream, Metronidazole Emulsion, Metronidazole Lotion, Brimonidine Tartrate Gel
* At least one medical record with a diagnosis code for rosacea (ICD-9: 695.3)
* At least 6 months of data history prior to the index date
* Had at least one encounter at the Reliant Medical Group within 3 months prior to 01 January 2015

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are using topical rosacea treatment
Sampling Method: Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2015-01-08 (Actual); Primary Completion 2016-03-10 (Actual); Study Completion 2016-03-10 (Actual)

PRIMARY OUTCOMES:
Self-reported concerns and importance of such concerns regarding their current topical rosacea treatments | Rosacea treatment in the past 4 weeks
  Assessed from the Rosacea Treatment Preference Questionnaire:
  Rated on a scale of 0 to 10, with 0 meaning not at all important and 10 meaning extremely important

SECONDARY OUTCOMES:
Self-reported likelihood of switching to a topical rosacea treatments | Rosacea treatment in the past 4 weeks
  Assessed from the Rosacea Treatment Preference Questionnaire:
  Rated on a scale of 0 to 10, with 0 meaning not at all likely and 10 meaning extremely likely
Quality of life | Rosacea treatment in the past 4 weeks
  Measured using Dermatology Life Quality Index (DLQI):
  The DLQI consists of 10 questions concerning symptoms and feelings, daily activities, leisure, work, and school, personal relationships and treatment
Treatment satisfaction | Rosacea treatment in the past 4 weeks
  Assessed by a score on the Treatment Satisfaction with Medicines Questionnaire (SATMED-Q). Scores will be standardized and expressed as a 0-100 standardized score
Self-reported concerns and importance (a rating scale) of such concerns that patients would consider when switching to a new topical rosacea treatment | Rosacea treatment in the past 4 weeks
  Extracted from the Rosacea Treatment Preference Questionnaire

OTHER OUTCOMES:
Baseline demographics and clinical characteristics: Age | Retrospective database analysis: encompassing patient data from up to 5 years
  Assessed from retrospective analysis of electronic medical records
Baseline demographics and clinical characteristics: Gender | Retrospective database analysis: encompassing patient data from up to 5 years
  Assessed from retrospective analysis of electronic medical records
Baseline demographics and clinical characteristics: Insurance type | Retrospective database analysis: encompassing patient data from up to 5 years
  Assessed from retrospective analysis of electronic medical records
Baseline demographics and clinical characteristics: Charlson Comorbidity Index (CCI) | Retrospective database analysis: encompassing patient data from up to 5 years
  Assessed from retrospective analysis of electronic medical records
Baseline demographics and clinical characteristics: Rosacea-relevant comorbidities and complications | Retrospective database analysis: encompassing patient data from up to 5 years
  Assessed from retrospective analysis of electronic medical records:
  Blepharitis (ICD-9: 373.0) Conjunctivitis (ICD-9: 372.0-372.2) Corneal neovascularization / keratitis (ICD-9: 370) Depression (ICD-9: 296.2-296.3) Migraine (ICD-9: 346)
Baseline demographics and clinical characteristics: Rosacea treatment-related adverse events | Retrospective database analysis: encompassing patient data from up to 5 years
  Assessed from retrospective analysis of electronic medical records:
  Burning/stinging/tingling (ICD-9: 782.0) Pruritus (ICD-9: 698) Scaling/dry skin/xerosis (ICD-9: 692.9, 706.8) Erythema/irritation (ICD-9: 695) Contact dermatitis (ICD-9: 692.3, 692.8, 692.9) Facial edema (ICD-9: 782.3) Acne (ICD-9: 706.1)
Current and past medication use | Retrospective database analysis: encompassing patient data from up to 5 years
  Assessed from retrospective analysis of electronic medical records
  Including:
  azelaic acid gel, azelaic acid cream, metronidazole gel, metronidazole cream, metronidazole lotion, metronidazole emulsion, brimonidine tartrate gel
Self-reported adverse events associated with patients' satisfaction/dissatisfaction | Rosacea treatment in the past 4 weeks
  Assessed from the Rosacea Treatment Preference Questionnaire:
  Rated on a scale of 0 to 10, with 0 meaning no pain/discomfort and 10 meaning unbearable pain/discomfort

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Boston, Massachusetts, United States